CLINICAL TRIAL: NCT02970357
Title: Evaluation of the Impact of a Therapeutic Education Program for Children With Type 1 Diabetes. A French Monocentric Prospective Study. Pilot Study
Brief Title: Evaluation of the Impact of a Therapeutic Education Program for Children With Type 1 Diabetes
Acronym: PROGETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GHRMSA 805; 2015-A017101-48 (Other: France: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2016-10-07; First posted 2016-11-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type I; Program Evaluation; Therapeutic Education; Children
Keywords: Evaluation; Therapeutic education; Type 1 Diabetes; Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enrolled patient (Other): Every patient of the Mulhouse Hospital with a type 1 diabetes who joins the study will be followed for 10 months. They will fill in the DIAPASON questionnaire and the quality of life WHO-5 questionnaire on the day of enrollment and 10 months after enrollment, at the end of the study. Young patients followed for a type 1 diabetes at the Mulhouse Hospital usually come every two months to see the pediatric endocrinologist, so the data collected for a regular visit will also be collected for the study every two months between the enrollment and the end of study participation.
  Interventions: Other: DIAPASON Questionnaire; Behavioral: WHO-5

INTERVENTIONS:
Other: DIAPASON Questionnaire — 50 item questionnaire of the French Youth Diabetes Association to evaluate one's theoretical knowledge about the diabetes disease. 6 main themes are evaluated :
  * what is diabetes
  * Monitoring
  * Hypoglycemia and Hyperglycemia
  * Nutrition
  * Insuline
Behavioral: WHO-5 — 5 item questionnaire of the World Health Organization about quality of life
  Other Names: Quality of Life Questionnaire

SUMMARY:
The needs of children and teens with type 1 diabetes are very specific and different from the adults with type 1 diabetes. Many organizations such as the World Health Organization or the International Society for Pediatric and Adolescent Diabetes, recommend a patient therapeutic education when it comes to children with type 1 diabetes.

This study aims to evaluate the impact of a therapeutic education program on theoretical knowledge of the disease and also on quality of life, on biological and clinical indicators.

DETAILED DESCRIPTION:
Structuring a therapeutic education program for patients with a chronic disease was the initiative of the French High Health Authority in June 2007.

The Prevention and Care of Pediatric Obesity and Pediatric Diabetes Organization of Mulhouse is a partner of the Mulhouse Hospital. Besides the usual care given at the hospital of Mulhouse for patients with a type 1 diabetes, both organizations also provide therapeutic education to these patients.

Each therapeutic education program is organized according to the patient's age. They can also be organized in a group or individually.

The aim of the therapeutic education is to help the young patients to cope with diabetes in their daily activities. Therapeutic education is known to bring good results for patients with diabetes, but there is no studies in France for children and teens with a type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment between January 15 to March 15, 2016
* Insulin-dependent type 1 Diabetes
* Treatment received at the Hospital of Mulhouse, France

Exclusion Criteria:

* Opposition to study participation
* Behavioral issues
* Uncontrolled psychological issue

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
The DIAPASON questionnaire | The outcome will be the change of the answers to the questionnaire from enrollment to the end of the study, ten months later.
  50 item questionnaire that evaluates the patient's theoretical knowledge of the type 1 diabetes disease. Questionnaire submitted to patients and a parent.

SECONDARY OUTCOMES:
Evolution of glycated hemoglobin | Throughout the study : on the enrollment day, 2 months after enrollment, 4 months after enrollment, 6 months after enrollment, 8 months after enrollment and 10 months after enrollment which is the end of the study participation
Occurrence of severe hypoglycemic events | Throughout the study : on the enrollment day, 2 months after enrollment, 4 months after enrollment, 6 months after enrollment, 8 months after enrollment and 10 months after enrollment which is the end of the study participation
Occurrence of ketoacidosis events | Throughout the study : on the enrollment day, 2 months after enrollment, 4 months after enrollment, 6 months after enrollment, 8 months after enrollment and 10 months after enrollment which is the end of the study participation
Need for care indicators | Throughout the study : on the enrollment day, 2 months after enrollment, 4 months after enrollment, 6 months after enrollment, 8 months after enrollment and 10 months after enrollment which is the end of the study participation
  Visits to the emergency room of a hospital, consultation with general practitioner
Behavioral indicators | Throughout the study : on the enrollment day, 2 months after enrollment, 4 months after enrollment, 6 months after enrollment, 8 months after enrollment and 10 months after enrollment which is the end of the study participation
  Evaluation of diabètes self-management, participation to therapeutic programs
Psychological indicators | On day 1, at enrollment, and 10months later, at the end of the study participation
  quality of life questionnaire for patient and parent

CONTACTS AND LOCATIONS:
Overall Officials: Fatiha GUEMAZI-KHEFFI, MD, Principal Investigator — Groupe Hospitalier de la Région de Mulhouse et Sud Alsace
Locations (1):
- GHRMSA, Mulhouse, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Study results — https://ecrin.app.unistra.fr/search/notice/view/ecrin-ori-72640